CLINICAL TRIAL: NCT01880879
Title: A Prospective Multicenter Trial Evaluating Helios Biodegradable Polymer Sirolimus-eluting Stent Safety and Effectiveness in Treatment of Coronary Artery Disease
Brief Title: A Prospective Multicenter Trial Evaluating Helios Biodegradable Polymer SES Safety and Effectiveness in CAD Treatment
Acronym: Pro-HOPE
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kinhely Bio-tech Co., Ltd. (Industry)
Collaborators: RenJi Hospital (Other); Peking University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro-HOPE
Record Dates: First submitted 2013-05-30; First posted 2013-06-19 (Estimated); Last update posted 2013-06-24 (Estimated); Status verified 2013-01

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery disease; PCI; stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- helios stent (Experimental): the group with helios stent implanted
  Interventions: Device: helios stent

INTERVENTIONS:
Device: helios stent — the group with helios stent implanted

SUMMARY:
research topic:helios After registration of clinical research bidders:kinhely bio-tech Co.Ltd study design:A prospective single treatment group multicenter clinical study Number of patients:Included in the subjects of 800 cases Main research purpose:Evaluation of safety and effectiveness Mainly studies the finish:1 year target lesion of the failure

Inclusion criteria :

one:Gender not limited at the age of 18 to 80 two:myocardial ischemia or angina symptoms of coronary artery disease three:A narrow is less than 50% treated with stents four:Comply with the instructions five:Voluntarily signed the informed consent form exclusion criteria: one:Pregnant women two:cardiac shock three:Against a suppository medicines or allergies four:Participated in other test research in the first 6 months five:Within 6 months after PCI plans to accept non cardiac surgery six:Non-compliant patient Follow-up time:A month for 6 months and 9 months to 1 year to 2 years follow-up progress plan:All center within 6 months after start of complete into the group

DETAILED DESCRIPTION:
no desired

ELIGIBILITY:
Inclusion Criteria:

* Any age 18 to 80 sex Myocardial ischemia or angina pectoris of coronary artery disease An application stents diameter stenosis greater than 50% Comply with the instructions Voluntarily signed the informed consent form

Exclusion Criteria:

* Pregnant women cardiac shock Intolerance to antithrombotic therapy or allergies 6 months prior to the start of the study involved in other studies Within 6 months after PCI plans to accept non cardiac surgery Non-compliant patient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2013-01; Primary Completion 2015-01 (Estimated); Study Completion 2015-01 (Estimated)

PRIMARY OUTCOMES:
1 year incidence of target lesion | 1year
  Target blood vessels caused by cardiac death and myocardial infarction and ischemia driven overall incidence of target lesion revascularization

SECONDARY OUTCOMES:
cardiac death Target blood vessels caused by myocardial infarction Ischemia driven target lesion revascularization of 1 year and 2 years,MACE, Stent thrombosis events,clinical success. | 2 years
  Death and myocardial infarction and thromboembolism events and hospitalizations and the incidence of major adverse cardiac events as the standard for safety evaluation
2 years, the incidence of various combination of the pathological changes of failure | 2 years
  Cardiac death drive target blood vessels lead to myocardial infarction and ischemia of the incidence of target lesion revascularization

OTHER OUTCOMES:
Rehospitalization rate | 2 years
  Stent placement in patients with the incidence of hospitalized again

CONTACTS AND LOCATIONS:
Locations (1):
- Yan chai hospital affiliated to Shanghai jiaotong university school of medicine, Shanghai, Shanghai Municipality, China